CLINICAL TRIAL: NCT03080753
Title: Treatment of Anal Incontinence Using Intersphincteric Implants (SphinKeeper)
Brief Title: Treatment of Anal Incontinence With Intersphincteric Implants
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study halted due to lower success rates than expected, after evaluation we have decided not to resume the study.
Sponsor: Region Skane (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Sphinkeeper 2017
Record Dates: First submitted 2017-03-06; First posted 2017-03-15 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Anal Incontinence; Fecal Incontinence
Keywords: Sphinkeeper; Intersphincteric implants; Gatekeeper
MeSH Terms: conditions — Encopresis; Fecal Incontinence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intersphincteric implants (Experimental): Treatment with intersphincteric implants in the anal sphincter using Sphinkeeper
  Interventions: Device: Sphinkeeper

INTERVENTIONS:
Device: Sphinkeeper — Intersphincteric implants in the anal sphincter
  Other Names: Gatekeeper; Intersphincteric implants

SUMMARY:
The purpose of this study is to determine whether treatment with intersphincteric implants is an effective and safe treatment option for patients with anal incontinence

DETAILED DESCRIPTION:
Treatment of anal incontinence (AI) remains a challenge - although conservative treatment can reduce the severity of many patients' AI, many continue to experience symptoms that severly affect their quality of life and ability to function properly both socially and professionally.

The level of AI is measured with the St Marks score (ranging from 0-24 where zero is complete continence).

Some patients with AI are shown to have defects in the anal sphincters (i.e. traumatic lesions post partum) and can be helped with reconstructive surgery. These procedures are effective but carry substantial risk for postoperative infection, and the healing process is painful.

One of the main treatment options for anal incontinence today is Sacral Nerve Stimulation (SNS), which is an effective but invasive and expensive treatment with a rather high level of infection. It is normally performed in two separate sessions and require life-long follow up and new surgical procedures every 6-7 years.

Historically artificial anal sphincters have been studied and shown to be effective but with high rates of infections leading to removal of the device. In more recent years studies have instead focused on "bulking agents" (injection of i.e. silicone in the submucosal space with the aim to increase the resting pressure of the anal canal), but the effect seems to be limited and the agents injected are rapidly resorbed by the body.

Treatment with intersphincteric implants is a novel treatment option for these patients. Available studies have shown good results regarding effect and a low frequence of postoperative infections. The implants rarely dislocate and are not resorbed by the body, which contributes to their long-term effectiveness. The operation is performed under a short general anaesthesia and in available studies the postoperative symptoms are few. The first technique described was called Gatekeeper (six implants), and this has since been completed by the Sphinkeeper (ten implants), which is the focus of the present study.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has been informed of the nature of the study, agrees to its provisions, and has provided written informed consent.
2. Subject must be at least 18 years of age
3. Subject must have a St Marks score of at least 11
4. Subject must be able to comply with study and study follow-up requirements.

Exclusion Criteria:

1. Subjects with Crohn's disease or Ulcerative colitis
2. Subject has (a history of) malignancy in the rectum or anal canal
3. Subject has an ongoing treatment with chemotherapy (all indications)
4. Subject has verified active anal fistula(e)
5. Subject is unable or unwilling to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-10-11 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2019-10-01 (Actual)

PRIMARY OUTCOMES:
Severity of anal incontinence | 12 months
  Reduction in St Marks score

SECONDARY OUTCOMES:
Postoperative infection | 12 months
  Rate of infection i.e. formation of abcess within the first year of treatment.
Change from baseline in pain scores on the VAS at 3 and 12 months. | Baseline, 3 months and 12 months
  VAS (Visual Analog Scale)

CONTACTS AND LOCATIONS:
Locations (1):
- Skåne University Hospital, Malmo, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ratto C, Parello A, Donisi L, Litta F, De Simone V, Spazzafumo L, Giordano P. Novel bulking agent for faecal incontinence. Br J Surg. 2011 Nov;98(11):1644-52. doi: 10.1002/bjs.7699. Epub 2011 Sep 16. PMID 21928378
- [Background] Ratto C, Buntzen S, Aigner F, Altomare DF, Heydari A, Donisi L, Lundby L, Parello A. Multicentre observational study of the Gatekeeper for faecal incontinence. Br J Surg. 2016 Feb;103(3):290-9. doi: 10.1002/bjs.10050. Epub 2015 Dec 1. PMID 26621029
- [Background] Ratto C, Donisi L, Litta F, Campenni P, Parello A. Implantation of SphinKeeper(TM): a new artificial anal sphincter. Tech Coloproctol. 2016 Jan;20(1):59-66. doi: 10.1007/s10151-015-1396-0. Epub 2015 Dec 12. PMID 26658726
- [Background] Al-Ozaibi L, Kazim Y, Hazim W, Al-Mazroui A, Al-Badri F. The Gatekeeper for fecal incontinence: Another trial and error. Int J Surg Case Rep. 2014;5(12):936-8. doi: 10.1016/j.ijscr.2014.08.002. Epub 2014 Oct 12. PMID 25460440
- [Background] Forte ML, Andrade KE, Lowry AC, Butler M, Bliss DZ, Kane RL. Systematic Review of Surgical Treatments for Fecal Incontinence. Dis Colon Rectum. 2016 May;59(5):443-69. doi: 10.1097/DCR.0000000000000594. PMID 27050607
- [Background] Thaha MA, Abukar AA, Thin NN, Ramsanahie A, Knowles CH. Sacral nerve stimulation for faecal incontinence and constipation in adults. Cochrane Database Syst Rev. 2015 Aug 24;2015(8):CD004464. doi: 10.1002/14651858.CD004464.pub3. PMID 26299888
- [Background] Maeda Y, Laurberg S, Norton C. Perianal injectable bulking agents as treatment for faecal incontinence in adults. Cochrane Database Syst Rev. 2013 Feb 28;2013(2):CD007959. doi: 10.1002/14651858.CD007959.pub3. PMID 23450581
- [Background] Norton C, Cody JD. Biofeedback and/or sphincter exercises for the treatment of faecal incontinence in adults. Cochrane Database Syst Rev. 2012 Jul 11;2012(7):CD002111. doi: 10.1002/14651858.CD002111.pub3. PMID 22786479
- [Background] Wang MH, Zhou Y, Zhao S, Luo Y. Challenges faced in the clinical application of artificial anal sphincters. J Zhejiang Univ Sci B. 2015 Sep;16(9):733-42. doi: 10.1631/jzus.B1400242. PMID 26365115